CLINICAL TRIAL: NCT02018146
Title: Cohort 2 Efficacy of Nasopharyngeal Ventilation With Endotracheal Tube for Patients With Predicted Difficult to Mask Ventilate
Brief Title: Cohort 2 Efficacy of Nasopharyngeal Ventilation With Endotracheal Tube for Surgery
Acronym: MASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rainer Lenhardt, Associate Professor, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 13.0570
Record Dates: First submitted 2013-10-29; First posted 2013-12-23 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: General Anesthesia With Endotracheal Intubation in Surgery
Keywords: Laryngeal Masks; Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasopharyngeal then mask (Other): Patients will be randomized to nasopharyngeal airway placement and ventilation followed by mask ventilation
  Interventions: Other: Nasopharyngeal then mask
- Mask then nasopharyngeal (Other): Patients will be randomized to mask ventilation followed by nasopharyngeal airway placement and ventilation
  Interventions: Other: Mask then nasopharyngeal

INTERVENTIONS:
Other: Mask then nasopharyngeal — Patients will be randomly assigned to Mask ventilation followed by naso-pharyngeal ventilation
  Arms: Mask then nasopharyngeal
Other: Nasopharyngeal then mask — Patients will be randomly assigned to naso-pharyngeal ventilation followed by mask ventilation.
  Arms: Nasopharyngeal then mask

SUMMARY:
Failed mask ventilation poses an increased risk of de-oxygenation to the patient undergoing general anesthesia. Nasopharyngeal ventilation may be a valid alternative for mask ventilation allowing for better oxygenation during the induction phase of general anesthesia. Oxygenation may be maintained better in case of difficult mask ventilation. This study evaluates this alternative method in comparison with the standard method of mask ventilation.

General Design This is a randomized, controlled, cross over study. Patients will be randomized to mask ventilation followed by nasopharyngeal airway placement and ventilation or vice versa.

Primary Study Endpoints We will test the hypothesis that ventilation via a nasally placed ETT is superior in its efficacy (as measured by tidal volume) to routine facemask ventilation in patients undergoing general anesthesia and endotracheal intubation for their surgery.

DETAILED DESCRIPTION:
General Design This is a randomized, controlled, cross over study. Patients will be randomized to mask ventilation followed by nasopharyngeal airway placement and ventilation or vice versa.

Primary Study Endpoints In cohort 2 we will test the hypothesis that ventilation via a nasally placed ETT is superior in its efficacy (as measured by tidal volume) to routine facemask ventilation in patients undergoing endotracheal intubation for general anesthesia. In cohort 1 the patient population was restricted to patients undergoing oto-laryngologic or oral maxillofacial surgery that required nasal intubation.

Subject Selection and Withdrawal General Characteristics of the Proposed Subject Population

Subjects will be enrolled at the University Pre-Op clinic or the University Pre-Op holding area. There is no data indicating that ethnicity affects airway management. We accordingly will accept patients from all minority groups. Based on the population of greater Louisville, we expect that 85% of the subjects will be Caucasian. We will include male and female patients in the study.

Anticipated Number of Research Subjects In cohort two we are planning to enroll 20 patients scheduled for endotracheal intubation and general anesthesia with their surgery. Patients will qualify for enrollment in the study if they meet the inclusion criteria as defined.

Inclusion Criteria

1. Subjects undergoing general anesthesia and require endotracheal intubation.
2. Adults patients 18 years or greater
3. Subjects are capable of understanding and signing the Informed Consent Form or have an acceptable representative capable of giving legally authorized consent on their behalf.
4. Meet three or more of predictive difficult to mask criteria as listed:

   1. Age = or > than 55
   2. BMI = or > than 30
   3. Edentulism
   4. History of snoring and/or a diagnoses of obstructive sleep apnea
   5. STOP/BANG score of three or greater
   6. Presesnce or a beard or mustach that covers the part of the face in conntact with the facemask edges
   7. Male gender
   8. History of neck radiation
   9. Mallampati score of III or IV

Exclusion Criteria I. Subjects will be excluded from this study in cases where there will not be an attempt at mask ventilation. This includes patients that will require an awake fiberoptic intubation as well as those needing a rapid sequence intubation.

II. Subjects with full stomachs, known hiatal hernia, and severe gastroesophageal reflux will be excluded.

III. Subjects with known or suspected basilar skull fractures will be excluded.

Subject Recruitment and Screening Subjects will be recruited by review of cases listed on the draft daily operating room schedule and schedule for pre-operative clinic at the University of Louisville hospital.

The study is confined to a short period at induction of anesthesia.

Visit 1 Screening Visit - at the screening visit subjects will undergo an airway exam.

Visit 2 Visit - Based on the screening results subject will be enrolled in to the study and randomized to one of the study groups. Immediately after randomization subject's nares will be prepped with two sprays of nasal decongestant bilaterally. NeoSynephrine nasal 0.5% spray will be used. Subject will be transferred to the OR.

Safety Assessments Routine anesthesia parameters (tidal volume, train of four, heart rate, oxygen saturation, end-tidal carbon dioxide, chest rise and BIS monitor) will be used to evaluate the safety of the proposed ventilation methods.

Effectiveness Assessments Tidal volume, train of four, heart rate, oxygen saturation, end-tidal carbon dioxide and chest rise will be used to evaluate the effectiveness of the study treatment Assessment of how difficult facemask ventilation actually was will use the method described by Warters(7). The Warters scale assigns points based on escalating levels of intervention necessary to ventilate the lungs. Additionally, the Warters scale accounts for situations in which a poor quality mask seal inhibits mask ventilation.

Sample Size Determination Preliminary data have shown that nasopharyngeal ventilation may improve applied tidal volumes compared to mask ventilation. Sample size analysis: a within-group difference of 50 ml tidal volume will be considered to be clinically significant in our study, because such difference will be equivalent to a 10% increase in tidal volume during naso-pharyngeal ventilation. Accordingly, per our a priori assessment, in order to detect an increase of 10% of tidal volume 16 patients will be required with 90% power at a significance level of 0.05. We propose to enroll 20 patients for this cross-over trial.

Statistical Methods Tidal volumes and airway pressures will be compared with paired T-tests. Data will be expressed as mean ± SD. Descriptive parameters and categorical variables will be compared using Chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing general anesthesia and require endotracheal intubation.
2. Adults patients 18 years or greater
3. Subjects are capable of understanding and signing the Informed Consent Form or have an acceptable representative capable of giving legally authorized consent on their behalf.
4. Meet three or more of predictive difficult to mask criteria as listed:

   1. Age = or > than 55
   2. BMI = or > than 30
   3. Edentulism
   4. History of snoring and/or a diagnoses of obstructive sleep apnea
   5. STOP/BANG score of three or greater
   6. Presesnce or a beard or mustach that covers the part of the face in conntact with the facemask edges
   7. Male gender
   8. History of neck radiation
   9. Mallampati score of III or IV

Exclusion Criteria:

* Subjects will be excluded from this study in cases where there will not be an attempt at mask ventilation. This includes patients that will require an awake fiberoptic intubation as well as those needing a rapid sequence intubation.
* Subjects with full stomachs, known hiatal hernia, and severe gastroesophageal reflux will be excluded.
* Subjects with known or suspected basilar skull fractures will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06; Primary Completion 2018-02-15 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 15 minutes
  After facemask or nasopharyngeal ventilation

SECONDARY OUTCOMES:
Airway pressure | 3 min after facemask or nasopharyngeal ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Background] Peterson GN, Domino KB, Caplan RA, Posner KL, Lee LA, Cheney FW. Management of the difficult airway: a closed claims analysis. Anesthesiology. 2005 Jul;103(1):33-9. doi: 10.1097/00000542-200507000-00009. PMID 15983454
- [Background] Domino KB, Posner KL, Caplan RA, Cheney FW. Airway injury during anesthesia: a closed claims analysis. Anesthesiology. 1999 Dec;91(6):1703-11. doi: 10.1097/00000542-199912000-00023. PMID 10598613
- [Background] Bund M, Walz R, Lobbes W, Seitz W. A tube in the pharynx for emergency ventilation. Acta Anaesthesiol Scand. 1997 Apr;41(4):529-30. doi: 10.1111/j.1399-6576.1997.tb04736.x. PMID 9150784
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Background] Han R, Tremper KK, Kheterpal S, O'Reilly M. Grading scale for mask ventilation. Anesthesiology. 2004 Jul;101(1):267. doi: 10.1097/00000542-200407000-00059. No abstract available. PMID 15220820
- [Background] Kheterpal S, Han R, Tremper KK, Shanks A, Tait AR, O'Reilly M, Ludwig TA. Incidence and predictors of difficult and impossible mask ventilation. Anesthesiology. 2006 Nov;105(5):885-91. doi: 10.1097/00000542-200611000-00007. PMID 17065880
- [Background] Warters RD, Szabo TA, Spinale FG, DeSantis SM, Reves JG. The effect of neuromuscular blockade on mask ventilation. Anaesthesia. 2011 Mar;66(3):163-7. doi: 10.1111/j.1365-2044.2010.06601.x. Epub 2011 Jan 25. PMID 21265818